CLINICAL TRIAL: NCT00703469
Title: A Phase I, Double-blind,Multicenter,Randomized,Placebo-controlled,Safety and Pharmacokinetic Dose-escalation Study of a Single Intravenous Administration of MDX-1106, a Fully Human Monoclonal Antibody to PD-1, in Subjects With Active Hepatitis C Genotype 1 Infection
Brief Title: A Study of MDX-1106 to Treat Patients With Hepatitis C Infection
Acronym: MDX1106-02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MDX1106-02; CA209-002 (Other: BMS)
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: Hepatitis C
Keywords: Hep C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MDX1106-02
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MDX1106-02 — Single dose
  Arms: 1
Drug: Placebo — Placebo single dose
  Arms: 2

SUMMARY:
This study examines the safety, tolerability, and immunogenicity of a single dose of MDX-1106 in patients with active hepatitis C genotype 1 or mixed hepatitis C genotype infection.

ELIGIBILITY:
Inclusion Criteria:

* Infection with hepatitis C genotype 1 or mixed hepatitis C genotype;
* Asymptomatic or nearly asymptomatic from hepatitis C;
* Previous therapy with interferon and ribavirin or peginterferon and ribavirin without an SVR or relapsed following an SVR;or Interferon naive subjects
* Chronically infected (at least 6 months since diagnosis) HCV-positive subjects;
* No evidence of bridging necrosis or cirrhosis;
* Liver biopsy within the last 2 years

Exclusion Criteria:

* Acute hepatitis C infection
* History of prior malignancy, acquired or inherited immunodeficiency or autoimmune disease either documented or anecdotal;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
safety, tolerability, and immunogenicity | One year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (7):
  - Advanced Clinical Resesarch Institute, Anaheim, California
  - Quest Clinical Research, San Francisco, California
  - Springfield Clinic Infectious Diseases, Springfield, Illinois
  - John Hopkins University School of Medicine, Viral Hepatitis Center, Baltimore, Maryland
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - The Liver Institute at Methodist Dallas, Dallas, Texas
  - Alamo Medical Research, San Antonio, Texas

REFERENCES:
- [Derived] Gardiner D, Lalezari J, Lawitz E, DiMicco M, Ghalib R, Reddy KR, Chang KM, Sulkowski M, Marro SO, Anderson J, He B, Kansra V, McPhee F, Wind-Rotolo M, Grasela D, Selby M, Korman AJ, Lowy I. A randomized, double-blind, placebo-controlled assessment of BMS-936558, a fully human monoclonal antibody to programmed death-1 (PD-1), in patients with chronic hepatitis C virus infection. PLoS One. 2013 May 22;8(5):e63818. doi: 10.1371/journal.pone.0063818. Print 2013. PMID 23717490